CLINICAL TRIAL: NCT02374359
Title: Atrial Tachycardia as a Predictor of Atrial Fibrillation, Stroke and Mortality in Cryptogenic Stroke
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Elisabet Pujol-Iglesias, Ph, Corporacion Parc Tauli
Other Study IDs: CPTCAR-EP201501
Record Dates: First submitted 2015-02-23; First posted 2015-02-27 (Estimated); Last update posted 2015-02-27 (Estimated); Status verified 2015-02

CONDITIONS: Cryptogenic Stroke; Atrial Fibrillation; Atrial Tachycardia
MeSH Terms: conditions — Ischemic Stroke; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- atrial tachycardia group: Patients diagnosed of cryptogenic stroke with atrial tachycardia in holter
  Interventions: Other: follow-up
- Non atrial tachycardia group (control group): Patients diagnosed of cryptogenic stroke with a normal holter
  Interventions: Other: follow-up

INTERVENTIONS:
Other: follow-up

SUMMARY:
There is few information about the association between supraventricular arrhythmia different from atrial fibrillation (AF) or atrial Flutter and the risk of stroke. In this study the investigators hypothesized that the presence of atrial tachycardia would lead to atrial fibrillation and recurrent stroke in patients hospitalized for cryptogenic stroke.

The investigators study the association of atrial tachycardia (AT), defined as four or more consecutive premature atrial beats, and AF, recurrent stroke and cardiovascular mortality in 192 consecutive patients hospitalized because of cryptogenic stroke. The follow-up was 12 months for all population

DETAILED DESCRIPTION:
The investigators review all consecutive patients that were hospitalized from stroke in our hospital (Neurology department) between January 2010 and September 2013, and who had the diagnosis of cryptogenic stroke at discharge. All patients routinely underwent 24-hour ECG recording and an echocardiography during the hospitalization. The investigators have a global population of 210 patients who met these characteristics.

The investigators analyze the presence of atrial tachycardia in 24-hour ECG register in patients with cryptogenic stroke. The investigators consider atrial tachycardia as four or more consecutive atrial ectopic beats.

The investigators analyze baseline characteristics (cardiovascular risk factors, renal function, left atrial size _measured in M mode echocardiography in long paraesternal axis_ and total number of premature atrial complexes in the 24-hour ECG monitoring.

The patients are stratified according to the presence or absence of atrial tachycardia in 24-hour ECG data.

The investigators follow the clinical events (AF, recurrent stroke or death) of patients from the electronical medical data of general physician and the re-hospitalizations for recurrent ictus in our hospital (which is the reference hospital of the zone) and mortality during 12 months.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients that were hospitalized from stroke in our hospital (Neurology department) between January 2010 and September 2013, and who had the diagnosis of cryptogenic stroke at discharge

Exclusion Criteria:

* Patients with non-cryptogenic stroke
* Patients with haemorragic stroke
* Patients with terminal disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We review all consecutive patients that were hospitalized from stroke in our hospital (Neurology department) between January 2010 and September 2013, and who had the diagnosis of cryptogenic stroke at discharge
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-02 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
ischemic stroke | 12 months

SECONDARY OUTCOMES:
atrial fibrillation | 12 months
cardiovascular mortality | 12 months
global mortality | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Corporacio Sanitaria Parc Tauli, Sabadell, Barcelona, Spain